CLINICAL TRIAL: NCT06572306
Title: Investigating the Impact of Pharmacist-led Flash Continuous Glucose Monitoring on Clinical and Behavioral Health Outcomes
Brief Title: Pharmacist-led Continuous Glucose Monitoring
Status: Recruiting | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kevin Cowart, Assistant Professor, University of South Florida
Other Study IDs: STUDY007451
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; endocrine disorders; continuous glucose monitor; pharmacist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Continuous glucose monitoring cohort (intervention): Freestyle libre 2 sensor devices will be used to monitor glucose. The sensors are worn on the upper arm and changed every 14 days. Each subject will have 5 visits with a pharmacist over 12 weeks. Subjects meeting inclusion criteria will include adults ≥18 years of age with type 2 diabetes and a hemoglobin A1c ≥ 8%. Subjects must have a compatible smartphone with the freestyle libre 2 sensor system. Subjects must have access to a glucometer to check blood glucose. Subjects must not have worn a continuous glucose monitor in the last 6 months to be eligible.
  Interventions: Device: FreeStyle Libre 2 Continuous Glucose Monitor
- Self-monitoring of blood glucose cohort (historical cohort): A retrospective chart review will be performed on patients seen by a clinic pharmacist between 1/1/2020-7/1/2024. Subjects in this group will include adults ≥18 years of age with type 2 diabetes and a hemoglobin A1c ≥ 8% and using a glucometer to monitor blood sugar. Exclusion criteria will be use of any continuous glucose monitoring device within the prior 6 months of the index date (defined as first visit with a pharmacist during study time frame).

INTERVENTIONS:
Device: FreeStyle Libre 2 Continuous Glucose Monitor — Subjects included in the intervention group (continuous glucose monitoring) will be recruited from the USF Health Department of Family Medicine. Each subject will be enrolled for 12 weeks.
  Groups: Continuous glucose monitoring cohort (intervention)

SUMMARY:
This is a pilot study. The goal of this prospective cohort study is to determine impact of pharmacist-led continuous glucose monitoring on glycemic control and health behavior change in people with type 2 diabetes. The main questions it aims to answer are:

1. to assess change in hemoglobin A1c in people with type 2 diabetes using continuous glucose monitoring under a pharmacist-led approach as compared to a pharmacist-led approach utilizing no continuous glucose monitoring (only self-monitoring blood glucose with a glucometer).
2. to assess change in continuous glucose monitoring-derived glycemic outcomes among the pharmacist-led continuous glucose monitoring cohort (intervention group)
3. to assess change in health behavior among the pharmacist-led continuous glucose monitoring cohort (intervention group)

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* hemoglobin A1c ≥ 8%
* compatible smartphone with FreeStyle Libre 2 continuous glucose monitoring system
* current use and access to a glucometer for self-monitoring of blood glucose

Exclusion Criteria:

* any continuous glucose monitor use within 6 months prior to study enrollment
* pregnant and planning to become pregnant during study time frame
* history of hypoglycemia requiring third party assistance
* history of diabetic ketoacidosis or hyperosmolar hyperglycemic state within 6 months prior to study enrollment
* known allergy to medical grade adhesives
* current use of systemic steroids for any medical condition
* current use of dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes with hemoglobin A1c ≥ 8%
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | Baseline to End of Study (12 weeks)
  Between-group difference in change in hemoglobin A1c at 12 weeks, %, compared between intervention and historical cohort

SECONDARY OUTCOMES:
Time in Range | Baseline to End of Study (12 weeks)
  Change in the time in range (70-180 mg/dL) at 12 weeks, %, compared within the intervention cohort
Mean Sensor Glucose | Baseline to End of Study (12 weeks)
  Change in mean sensor glucose concentration at 12 weeks, mg/dL, compared within the intervention cohort
Time Below Range | Baseline to End of Study (12 weeks)
  Change in time below range (< 54mg/dL and < 70 mg/dL) at 12 weeks, %, compared within the intervention cohort
Time Above Range | Baseline to End of Study (12 weeks)
  Change in time above range (> 180 mg/dL and > 250 mg/dL) at 12 weeks, %, compared within the intervention cohort
Glycemic Variability | Baseline to End of Study (12 weeks)
  Change in glycemic variability (standard deviation, and Coefficient of variance) at 12 weeks, compared within the intervention cohort
Time in Range Increase 5% | Baseline to End of Study (12 weeks)
  Change in the number of subjects increasing 5% or more in time in range (70-180 mg/dL) at 12 weeks, compared within the intervention cohort
Time in Range Increase 10% | Baseline to End of Study (12 weeks)
  Change in the number of subjects increasing 10% or more in time in range (70-180 mg/dL) at 12 weeks, compared within the intervention cohort
>70% Time in Range | Baseline to End of Study (12 weeks)
  Change in the number of subjects achieving > 70% time in range (70-180 mg/dL) at 12 weeks, compared within the intervention cohort
Hemoglobin A1c <7% | Baseline to End of Study (12 weeks)
  Change in the number of subjects achieving hemoglobin A1c < 7% at 12 weeks compared between intervention and historical cohort
Hemoglobin A1c <8% | Baseline to End of Study (12 weeks)
  Change in the number of subjects achieving hemoglobin A1c < 8% at 12 weeks compared between intervention and historical cohort
Summary of Diabetes Self-Care Activities Measure | Baseline to End of Study (12 weeks)
  Change in the Summary of Diabetes Self-Care Activities Measure at 12 weeks, compared within the intervention group. Scored on an 8-point likert scale (0-7). Higher scores indicate better compliance with diabetes self-care, whereas a lower score indicate poor self-care performance.
Continuous Glucose Monitoring Survey Responses | Baseline to End of Study (12 weeks)
  Change in survey responses at 12 weeks, compared within the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cowart, PharmD, MPH, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - USF Health Department of Family Medicine - Morsani Center for Advanced Health Care, Tampa, Florida
  - USF Health Department of Family Medicine - University Partnership Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowart K, White RT, Olson K, Carris NW, Hanna K, Zgibor J. Impact of Pharmacist-Led Continuous Glucose Monitoring on Clinical Outcomes in People With Type 2 Diabetes in Primary Care: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2025 May 23;14:e67014. doi: 10.2196/67014. PMID 40409747